CLINICAL TRIAL: NCT00084045
Title: Mother Infant Rapid Intervention at Delivery (MIRIAD)
Brief Title: Voluntary HIV Counseling, Testing, and Medication for Pregnant Women to Prevent Mother-to-Child HIV Transmission
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PACTG P1031A; MIRIAD
Record Dates: First submitted 2004-06-04; First posted 2004-06-07 (Estimated); Last update posted 2012-10-30 (Estimated); Status verified 2012-10

CONDITIONS: HIV Infections
Keywords: HIV Seronegativity; Treatment Naive; Pediatric HIV; Perinatal Transmission
MeSH Terms: conditions — HIV Infections

INTERVENTIONS:
Procedure: Intrapartum HIV counseling/testing
Procedure: Postpartum HIV counseling/testing

SUMMARY:
Voluntary HIV counseling and testing (VCT) and anti-HIV drugs for pregnant women and their newborns decrease rates of mother-to-child transmission (MTCT) of HIV. This study will determine the acceptability of HIV counseling and rapid testing prior to delivery and will compare the usefulness of VCT prior to birth versus after birth in preventing MTCT of HIV in pregnant women in Cape Town, South Africa. This study will also determine the acceptability and effectiveness of giving anti-HIV medications to prevent MTCT of HIV.

DETAILED DESCRIPTION:
Pediatric HIV infection is a major public health problem in South Africa, and is primarily caused by MTCT of HIV. Strategies to prevent MTCT have been successfully employed when a mother's HIV status is known. However, there is concern in South Africa that it is unethical to offer HIV testing to women in the intrapartum period when they are experiencing the physical and emotional stress of labor. This study will compare the acceptability and accuracy of intrapartum and postpartum VCT in pregnant women of unknown HIV status in Cape Town, South Africa.

Pregnant women of unknown HIV status coming to a participating hospital to deliver will be asked to enter the trial. Women will be assigned to either intrapartum or postpartum VCT depending on the week during which they come to the hospital. The intervention (intrapartum or postpartum VCT) for the week will be randomly assigned and all women enrolling in the trial in a given week will receive the same intervention.

All women will receive HIV counseling prior to testing. Women in the intrapartum VCT group who are HIV infected will receive antiretrovirals (ARV) prior to delivery to prevent MTCT, and their infants will receive ARV within 3 days of birth. Infants born to HIV infected women in the postpartum VCT group will receive ARV as soon as possible after confirmation of the mother's positive test. All women will receive post-test counseling prior to discharge.

HIV VCT, medical history assessment, and physical exam will occur at study entry. A small subset of both HIV infected and uninfected mothers will be asked for their opinions regarding peripartum HIV VCT and MTCT prevention strategies during qualitative assessments.

Infants will undergo physical exam within 2 days of birth, medical history assessment within 2 days of birth and at 3 additional times between 6 and 14 weeks of age, and HIV testing within 2 days of birth and at 2 additional times between 6 and 12 weeks of age.

ELIGIBILITY:
Inclusion Criteria for Women:

* Unknown HIV infection status
* At least seven months pregnant
* Women in active labor who have planned induction or Caesarean delivery or any other condition requiring planned delivery

Inclusion Criteria for Infants:

* Mother is participating in study
* Mother is HIV infected

Exclusion Criteria for Women:

* Women in labor who need immediate delivery
* Obstetrical emergencies in which the woman is medically unstable or requires emergency delivery
* Diagnosed fetal death or fetal condition requiring abortion

Min Age: 14 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 283 (Actual)
Dates: Start 2004-11; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Time required to obtain informed consent
time from initiation of HIV pre-test counseling until test results are available
proportion of test evaluations completed before delivery
proportion of test evaluations completed before hospital discharge
proportion of women who agree to HIV testing
proportion of women identified as HIV infected during labor who accept ARV prophylaxis
proportion of women identified as HIV infected after birth who accept ARV therapy for their infants
timing of infant ARV prophylaxis initiation after birth, as a proportion of infants born to women identified as HIV infected after birth and as a continuous variable
timing of mother ARV initiation as a proportion of women identified as HIV infected during labor and as a continuous variable
qualitative measures (defined as available space, study staff allocation, support for counseling and testing, and women's perceptions and opinions of counseling and testing)

SECONDARY OUTCOMES:
Proportion of women with undocumented HIV infection who are tested and determined to be HIV infected peripartum
performance of rapid HIV tests as measured by sensitivity and specificity
proportion of infants who complete the Week 6 study visit and efforts needed to accomplish this visit
proportion of infants being fed according to the method chosen at discharge (defined as exclusive breastfeeding, exclusive formula feeding, or mixed feeding), as reported by the mother at Week 6
proportion of HIV-exposed infants who acquire HIV infection during delivery and after birth
acceptance of HIV counseling and testing among clinical personnel at primary, secondary, and tertiary care facilities

CONTACTS AND LOCATIONS:
Overall Officials: Robert Maupin, Jr., MD, Study Chair — Louisiana State University Health Science Center; Mitchell Besser, MD, Study Chair — Department of Obstetrics and Gynecology, Groote Schuur Hospital Observatory
Locations (2):
- South Africa (2):
  - Hottentots Holland Hospital, Cape Town
  - Maccassar Community Health Clinic, Cape Town

REFERENCES:
- [Background] Leroy V, Sakarovitch C, Cortina-Borja M, McIntyre J, Coovadia H, Dabis F, Newell ML, Saba J, Gray G, Ndugwa Ch, Kilewo Ch, Massawe A, Kituuka P, Okong P, Grulich A, von Briesen H, Goudsmit J, Biberfeld G, Haverkamp G, Weverling GJ, Lange JM; Ghent Group on HIV in Women and Children. Is there a difference in the efficacy of peripartum antiretroviral regimens in reducing mother-to-child transmission of HIV in Africa? AIDS. 2005 Nov 4;19(16):1865-75. doi: 10.1097/01.aids.0000188423.02786.55. PMID 16227795
- [Background] McIntyre J. Strategies to prevent mother-to-child transmission of HIV. Curr Opin Infect Dis. 2006 Feb;19(1):33-8. doi: 10.1097/01.qco.0000200290.99790.72. PMID 16374215
- [Background] Newell ML. Current issues in the prevention of mother-to-child transmission of HIV-1 infection. Trans R Soc Trop Med Hyg. 2006 Jan;100(1):1-5. doi: 10.1016/j.trstmh.2005.05.012. Epub 2005 Oct 7. PMID 16214193
- [Result] Bulterys M, Jamieson DJ, O'Sullivan MJ, Cohen MH, Maupin R, Nesheim S, Webber MP, Van Dyke R, Wiener J, Branson BM; Mother-Infant Rapid Intervention At Delivery (MIRIAD) Study Group. Rapid HIV-1 testing during labor: a multicenter study. JAMA. 2004 Jul 14;292(2):219-23. doi: 10.1001/jama.292.2.219. PMID 15249571
- [Result] Jamieson DJ, O'Sullivan MJ, Maupin R, Cohen M, Webber MP, Nesheim S, Lampe M, Garcia P, Lindsay M, Bulterys M. The challenges of informed consent for rapid HIV testing in labor. J Womens Health (Larchmt). 2003 Nov;12(9):889-95. doi: 10.1089/154099903770948113. PMID 14670168